CLINICAL TRIAL: NCT01814241
Title: Mechanisms of Desensitization During Peanut Oral Immunotherapy
Acronym: PnOIT4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-0900; R01AI068074 (NIH)
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2017-03

CONDITIONS: Food Hypersensitivity
Keywords: Peanut allergy
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label peanut OIT (Experimental): Open label orally ingested peanut flour with maintenance dose of 1450mg
  Interventions: Drug: Open label peanut OIT

INTERVENTIONS:
Drug: Open label peanut OIT — Subject will take increasing amounts of peanut protein up to a maximum maintenace dose of 1450mg.
  Other Names: Peanut flour

SUMMARY:
The purpose of this study is to attempt to understand how desensitization works in peanut allergic children who are undergoing oral immunotherapy (OIT) to peanut. We want to identify the early changes in the desensitization process the immune cells undergo to become desensitized to the peanut protein.

DETAILED DESCRIPTION:
Peanut allergic children will undergo an oral food challenge (OFC) to 1 gm peanut protein in order to accomplish two objectives: (1)to confirm the diagnosis of peanut allergy, and (2) to measure the amount of peanut protein it takes to cause an allergic reaction. Each subject will then undergo a modified rush phase in which the subject receives 6 doses of peanut protein in one day. The build-up phase begins afterward in which the subject's dose of peanut protein is increased every 2 weeks for 36 weeks. After the final build-up dose, the subject consumes that dose for 2 weeks after which he or she returns to the food allergy center for the second food challenge. If the subject successfully consumes this food challenge without symptoms, the daily dosing of peanut protein will be stopped and the subject will then undergo a third food challenge. If the subject successfully consumes the peanut protein during that challenge, he or she will return for a fourth food challenge to peanut.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to up to 12 years of age of any gender, race, or ethnicity.
* Minimum weight 16 kg at the time of enrollment.
* Physician diagnosis of peanut allergy OR convincing clinical history of an allergic reaction to peanut.
* Detectable serum peanut -specific IgE level (CAP-FEIA ≥ 0.35 kU/L) and a positive SPT (wheal ≥ 3mm on skin prick test to peanut extract compared to a negative control.)
* Allergic reaction to ≤ 1 gm peanut protein during a blinded oral challenge test conducted at screening (e.g., a double-blinded, placebo-controlled food challenge [DBPCFC]).
* Written informed consent from parent/guardian.
* Written assent from subject if applicable
* Consumption of oat-containing product within 90 days prior to enrollment

Exclusion Criteria:

* History of allergic reaction to peanut consistent with severe anaphylaxis (defined as hypotension/shock; or neurologic impairment).
* Chronic disease other than asthma, atopic dermatitis, rhinitis requiring therapy; e.g., heart disease or diabetes.
* Active eosinophilic gastrointestinal disease in the past 2 years
* Participation in any interventional study for the treatment of food allergy in the 6 months prior to visit -1
* Inhalant allergen immunotherapy that has not yet reached maintenance dosing.
* Asthma defined as moderate or severe persistent by National Asthma Education and Prevention Program Expert Panel Guidelines (e.g. asthma that requires more than fluticasone 440 mcg or its equivalent daily for adequate control).
* Inability to discontinue antihistamines for skin testing, OFC and the initial dose escalation.
* Use of omalizumab or other non-traditional forms of allergen immunotherapy (e.g., oral or sublingual) in the 12 months prior to visit -1.
* Any systemic therapy which in the judgment of the investigator could be immunomodulatory (e.g. rituximab) in the 12 months prior to visit -1, Systemic corticosteroid therapy of up to a total of three weeks is allowed.
* Use of investigational drug in 90 days prior to visit -1.
* Plan to use any investigational drug during the study period.
* The presence of any medical condition that the investigator deems incompatible with participation in the trial.
* Inability to speak English.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Burks, MD, Principal Investigator — UNC Chapel Hill; Edwin Kim, MD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label Peanut OIT
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 8.8 [5.9 to 11.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Develop Desensitization
Description: The percentage of peanut allergic subjects who develop desensitization as defined by being able to consume 5000mg of peanut protein during a double blind food challenge after completing a build-up phase of peanut OIT.
Time Frame: 40 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 16
percentage of participants | 81.25

2. Secondary Outcome: Percentage of Subjects Who Maintain Desensitization Once OIT is Stopped
Description: The percentage of subjects who maintain desensitization once the OIT is withdrawn at 1, 2, 3, and 4 week intervals.
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 14
percentage of participants | 21.43

3. Other Pre Specified Outcome: Change From Baseline in the Wheal Diameter, as Assessed by the Skin Prick Test (SPT) to Peanut
Description: Allergic reactivity of mast cells is assessed by skin prick testing through measurement of the wheal diameter after exposure to peanut. This outcome measure reports the change in skin prick test wheal diameter from baseline through the end of the treatment period.
Time Frame: 44 weeks
Measure: Mean (Full Range); unit: mm
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 16
mm | -8.8 [-24.5 to 5.5]

4. Other Pre Specified Outcome: Change in Peanut Specific Immunoglobin E (IgE) From Baseline Until Desensitization Food Challenge
Description: The investigation of mechanistic changes that occur in the immune system over the duration of the study - Peanut specific immunoglobin E (IgE)
Time Frame: 44 weeks
Population: Blood work was not able to be obtained from 1 of 16 evaluable subjects
Measure: Median (Full Range); unit: kU/L of peanut-specific IgE
Groups:
- Open Label Peanut OIT: Subject cohort receiving open label orally ingested peanut flour with maintenance dose of 1450mg
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 15
kU/L of peanut-specific IgE | -19 [-466 to 544.5]

5. Other Pre Specified Outcome: Change in Immunoglobin G4 (IgG4) to Peanut From Baseline Until Desensitization Food Challenge
Description: The investigation of mechanistic changes that occur in the immune system dover the duration of the study - Immunoglobin G4 (IgG4) to peanut
Time Frame: 44 weeks
Population: Blood work was not able to be obtained from 1 of 16 evaluable subjects
Measure: Median (Full Range); unit: mg/dL of IgG4
Arm/Group | Open Label Peanut OIT
Number analyzed (Participants) | 15
mg/dL of IgG4 | 3.68 [0.47 to 92.88]

ADVERSE EVENTS:
Time Frame: 31 months
Arm/Group | Open Label Peanut OIT
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 15/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Peanut OIT (N=20)
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Erythematous rash (Skin and subcutaneous tissue disorders) | 4
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal itching (Skin and subcutaneous tissue disorders) | 7
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0
Itchy nose (Skin and subcutaneous tissue disorders) | 1
Skin itch (Skin and subcutaneous tissue disorders) | 2
Lip or eye swelling (Skin and subcutaneous tissue disorders) | 4
Eye itch (Eye disorders) | 1
Eye tearing (Eye disorders) | 0
Hives (Skin and subcutaneous tissue disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0
Throat tightness (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No